CLINICAL TRIAL: NCT00476203
Title: Effect of Yoga on Weight and Fatigue in Breast Cancer Patients Study
Brief Title: Yoga Study in Breast Cancer Patients
Acronym: Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Mark Boyer, Director of Sponsored Research, Fred Hutchinson Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHS - 6434; U54CA116847-01 (NIH)
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Yoga; Quality of Life; Obesity; Fatigue; Weight
MeSH Terms: conditions — Breast Neoplasms; Obesity; Fatigue; Body Weight | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Immediate yoga classes offered
  Interventions: Behavioral: Yoga
- 2 (Other): Delayed yoga classes (after 6 months) offered [wait list control group]
  Interventions: Other: Delayed yoga classes

INTERVENTIONS:
Behavioral: Yoga — Instructor-led yoga classes 1/time per week + 4 days of home practice
  Arms: 1
Other: Delayed yoga classes — Delayed yoga classes (after 6 months) offered [wait list control group]
  Arms: 2

SUMMARY:
This purpose of this study is to test whether a 6-month yoga program improves quality of life and reduces fatigue and weight gain in breast cancer survivors.

DETAILED DESCRIPTION:
Women who are overweight or obese have a higher risk of breast cancer than normal weight women. Furthermore, women who are overweight or obese or gain weight after diagnosis have an increased risk of recurrence or dying from breast cancer compared with normal weight women. Yoga has been associated with reduced weight gain and weight loss in persons without cancer. However, no studies have tested whether yoga leads to less weight gain or weight loss in breast cancer patients. Both obesity and the sequelae of breast cancer therapy can result in reduced health-related quality of life and severe fatigue, which may also be favorably affected by yoga practice. The specific aims of the proposed trial are to examine, in women with Stage 0-IIIa breast cancer who are at least 3 months post primary treatment for their disease (other than tamoxifen or aromatase inhibitors), the effects of a 6-month yoga intervention on health-related quality of life, fatigue, and body weight.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 21-75
* Diagnosed with a primary breast cancer Stage 0-IIIa
* Current tamoxifen or aromatase inhibitor use is allowed
* At least 3 months post treatment (e.g., surgery, chemotherapy, or radiation therapy)
* BMI: 24 kg/m2 or greater (If Asian or Asian-American BMI: 23 kg/m2 or greater)
* No contraindications to participating in a yoga program
* Able to come for clinic visits, and attend weekly classes, and fill out questionnaires and logs in English
* Gives informed consent, agrees to be randomly assigned

Exclusion Criteria:

* Plans to leave the study area within the follow-up period
* Is pregnant or plans to become pregnant during the study period.
* History of myocardial infarction (heart attack) or stroke in the previous 6 months, or diabetes (current diagnosis)
* Has practiced yoga more than 1 time per month in the past six months.
* Current use of medications likely to interfere with adherence to interventions or study outcomes
* Alcohol or drug abuse, significant mental illness (as assessed by study staff impression)

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-05; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
quality of life, fatigue, and body weight | baseline, 6 months, 12 months

SECONDARY OUTCOMES:
waist and hip circumference | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alyson Littman, PhD, Study Director — Department of Epidemiology, UW; Anne McTiernan, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Result] Littman AJ, Bertram LC, Ceballos R, Ulrich CM, Ramaprasad J, McGregor B, McTiernan A. Randomized controlled pilot trial of yoga in overweight and obese breast cancer survivors: effects on quality of life and anthropometric measures. Support Care Cancer. 2012 Feb;20(2):267-77. doi: 10.1007/s00520-010-1066-8. Epub 2011 Jan 5. PMID 21207071